CLINICAL TRIAL: NCT07008404
Title: A Pilot Study to Assess the Feasibility of an Online Cognitive Behavioural Therapy Application (Mahana IBS™, Mahana Therapeutics) in the Management of Irritable Bowel Syndrome
Brief Title: Feasibility of an Online Cognitive Behavioural Therapy Application (Mahana IBS™, Mahana Therapeutics) in the Management of Irritable Bowel Syndrome
Acronym: MahanaPilot
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Producer decided to stop commercialization of the Mahana app
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23GA006; IRAS number: 325405 (Other: IRAS)
Record Dates: First submitted 2025-06-03; First posted 2025-06-06 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Irritable Bowel Syndrome (IBS)
Keywords: CBT; pilot study
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CBT (Other): online cognitive behavioral therapy
  Interventions: Device: online cognitive behavioral therapy

INTERVENTIONS:
Device: online cognitive behavioral therapy — unguided online cognitive behavioral therapy app

SUMMARY:
Irritable bowel syndrome (IBS) is a very common condition where patients suffer from recurrent episodes of tummy pain associated with the way the bowel works (either constipation, diarrhoea, or a mix of both). The cause of this condition is still unclear, but it has been shown that, for some people their bowel is more sensitive to normal things like meals and stress. Studies have confirmed that psychological therapies are helpful for IBS. Cognitive behavioural therapy (CBT) has been shown to be one of the most helpful over the long term. CBT is a type of talking therapy that helps patients to examine their thoughts, feelings, and behaviours, with a view to change some of them. CBT can help patients to influence their physical IBS symptoms with the help of this therapy. The National Institute for Health and Care Excellence (NICE) recommends CBT in patients who not respond to medications and experience ongoing symptoms. A recent large study conducted in UK has demonstrated that an online version of this CBT, delivered with the help of a therapist, was effective in treating symptoms of IBS. However, in the UK, there is a lack of therapists to support the online version.

A small study conducted in USA has demonstrated that an unguided version of this online CBT (called Mahana IBS) could be as effective as the therapist guided one. This study was small and only enrolled patients who self-referred. This does not reflect what normally happens in clinical practice where patients are normally proposed a treatment by a clinician.

There is a plan tu run a multicentre study in the UK to show that Mahana IBS works (as a mobile/tablet app) for patients with IBS, in clinical practice. Before running this study, it is necessary to get some experience of its use. So, in this pilot study, the aim is to find out if it is feasible to use this CBT app in real-world clinical practice in UK, and whether this improves IBS symptoms and mental health status. In particular the aim is to understanding whether UK patients normally seen in hospital are interested in using this CBT app, can use and complete the planned CBT course, and whether this helps them improving their IBS symptoms and mental health status. Patients will be recruited from Nottingham University Hospital Trust, and the plan is to recruit 60 patients with a diagnosis of IBS.

DETAILED DESCRIPTION:
In this pilot study, the aim is to include IBS patients as would be typically encountered in real-world, UK healthcare settings to evaluate the response to the unguided Mahana IBS™, Mahana Therapeutics app-based CBT application for the management of IBS. The results of this pilot study would provide the basis to conduct a feasibility randomised-controlled trial in secondary care settings to evaluate the current barriers/facilitators to the use of Mahana IBS™ in the real-world clinical practice, as well as obtain information to decide the primary endpoint to be used in a definitive randomised controlled, cost-effectiveness trial comparing the use the app (experimental arm) vs. a treatment as usual (control arm). This study would also provide data on the resources required, including the necessary study time scale;

ELIGIBILITY:
Inclusion Criteria:

* Patients capable of giving informed consent
* Older than 18 years of age
* Patients referred by their GP to secondary/tertiary care with clinical symptoms of IBS (as per NICE guidelines)
* Have regular access to a device with internet

Exclusion Criteria:

* Patients with concurrent organic gastrointestinal disease (inflammatory bowel disease, coeliac disease, cancer)
* Concurrent major confounding condition, e.g., alcohol or substance abuse in the last 2 years (clinician's judgement)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male and female
Enrollment: 20 (Actual)
Dates: Start 2024-01-17 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
retention rate of patients provided with the Mahana IBS™ application | from enrollment to end of treatment at 12 weeks
  number of patients completing the entire course of the treatment

SECONDARY OUTCOMES:
change in the IBS symptom severity scale score for patients | From enrollment to the end of treatment at 12 weeks
  difference between score at baseline and at the end of treatment, scale from 0 to 500, where 500 means worse score
change in the generalised anxiety and depression score-7 | rom enrollment to the end of treatment at 12 weeks
  difference between the score at baseline and at the end of the treatment, scale from 0 to 21, where 21 means worse score
change in the patient health questionnaire-9 score | From enrollment to the end of treatment at 12 weeks
  difference in score between baseline and end of the treatment, scale from 0 to 27, where 27 means worse score

CONTACTS AND LOCATIONS:
Locations (1):
- Translational Medical Sciences, Nottingham, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Access Criteria: after publication

REFERENCES:
- [Background] Gerstein HC, Sattar N, Rosenstock J, Ramasundarahettige C, Pratley R, Lopes RD, Lam CSP, Khurmi NS, Heenan L, Del Prato S, Dyal L, Branch K; AMPLITUDE-O Trial Investigators. Cardiovascular and Renal Outcomes with Efpeglenatide in Type 2 Diabetes. N Engl J Med. 2021 Sep 2;385(10):896-907. doi: 10.1056/NEJMoa2108269. Epub 2021 Jun 28. PMID 34215025
- [Background] Everitt H, Moss-Morris R, Sibelli A, Tapp L, Coleman N, Yardley L, Smith P, Little P. Management of irritable bowel syndrome in primary care: the results of an exploratory randomised controlled trial of mebeverine, methylcellulose, placebo and a self-management website. BMC Gastroenterol. 2013 Apr 21;13:68. doi: 10.1186/1471-230X-13-68. PMID 23602047